CLINICAL TRIAL: NCT06644573
Title: Evaluating the Efficacy and Safety of PROSOMNIA Sleep Therapy™ in Patients With Sleep Deprivation and Chronic Insomnia
Acronym: PSHW
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nyree Penn (Industry)
Collaborators: Masimo Corporation (Industry); PROSOMNIA Sleep Health & Wellness (Industry)
Responsible Party: Sponsor-Investigator, Nyree Penn, MHSc., CEO, PROSOMNIA Sleep Health & Wellness
Organization: PROSOMNIA Sleep Health & Wellness (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROSOMNIAsleep
Record Dates: First submitted 2024-09-08; First posted 2024-10-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia; Sleep Deprivation; REM Behavior Disorder; REM Sleep Behavior Disorder; REM Sleep Measurement; Insomnia; Insomnia Related to Specified Disorder; Insomnia Due to Other Mental Disorder; Insomnia Comorbid to Psychiatric Disorder; Insomnia Due to Anxiety and Fear; Insomnia Related to Another Mental Condition; Insomnia Disorders; Idiopathic Hypersomnia; Sleep Disorders, Circadian Rhythm; Post Trauma Nightmares; PTSD - Post Traumatic Stress Disorder; Sleep Quality; Anesthesia; Anxiety; Depression; Mental Health; Alzheimer Disease or Associated Disorder; Parkinsons; Circadian Rhythm; Circadian Dysregulation; PTSD; Post-Traumatic; Post-Traumatic Stress Disorder Complex; Military Combat Stress Reaction; Sleep; Military Activity; Veterans; Shift Work Sleep Disorder; Menopause Related Conditions; Pain; Cancer Pain; Athletes
Keywords: SLEEP; PROSOMNIA Sleep; PROSOMNIA Sleep Therapy; PSTx; PROSOMNIA; Anesthesia Sleep; REM Sleep; REM Sleep Therapy; PROSOMNIA Sleep Health; PROSOMNIA Sleep Wellness; PROSOMNIA Sleep Treatment; Nyree; Nyree Penn; Propofol; Propofol Sleep; Diprivan; Diprivan Sleep; PROSOMNIA Sleep Health and Wellness; Insomnia; Sleep Deprivation; IH; Idiopathic Hypersomnia; Sleep Debt; PTSD; Mental Health; Anxiety; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation; REM Sleep Behavior Disorder; Idiopathic Hypersomnia; Sleep Disorders, Circadian Rhythm; Combat Disorders; Anxiety Disorders; Depression; Psychological Well-Being; Alzheimer Disease; Chronobiology Disorders; Stress Disorders, Post-Traumatic; Pain; Cancer Pain | interventions — Propofol; Electroencephalography

STUDY DESIGN:
Intervention Model Description: This clinical trial follows a Single Group Assignment model, where all enrolled participants receive the same intervention-PROSOMNIA Sleep Therapy (PSTx). The model is open-label, meaning both the participants and researchers are aware of the treatment being administered. There is no placebo or control group in this trial, as the focus is to directly evaluate the safety and efficacy of PSTx for chronic insomnia and related REM sleep disorders.
  The intervention involves the use of monitored anesthesia care (MAC) to induce and regulate REM sleep, using Diprivan/Propofol under the supervision of an Anesthesiologist and a Certified Anesthetist. Continuous EEG monitoring ensures proper sleep architecture is achieved during the therapy session, and adjustments are made in real-time to optimize therapeutic outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-Arm - PROSOMNIA Sleep Therapy (Experimental): Description: All eligible participants in this study will be assigned to a single arm and receive the same intervention, PROSOMNIA Sleep Therapy. This involves a controlled, anesthesia-induced sleep session using Diprivan/Propofol, administered under the supervision of an Anesthesiologist. Monitoring will include American Society of Anesthesiologists (ASA) standard monitoring and real-time EEG to track sleep stages and brain activity during the procedure.
  Interventions: PROSOMNIA Sleep Therapy, involving the administration of Diprivan/Propofol, a FDA-approved anesthetic, to induce sleep in individuals with chronic insomnia, sleep deprivation and/or REM sleep disparities. This treatment is intended to reduce sleep pressure, decrease sleep onset latency, enhance REM sleep duration, and improve overall sleep quality. Continuous EEG monitoring to track sleep architecture and blood serum uric acid tests to identify adenosine release.
  Interventions: Procedure: PROSOMNIA Sleep Therapy™ (PSTx); Procedure: Anesthesia-Induced Sleep Therapy; Drug: Diprivan (propofol), Astra-Zeneca; Device: Continuous EEG Monitoring

INTERVENTIONS:
Procedure: PROSOMNIA Sleep Therapy™ (PSTx) — PROSOMNIA Sleep Therapy (PSTx) is a novel intervention designed to manage homeostatic sleep pressure by leveraging an anesthesia-induced protocol. Using Diprivan/Propofol, PSTx rapidly induces REM sleep, clearing adenosine from the brain and reducing sleep pressure more efficiently than traditional methods. Monitored in real-time via EEG, this therapy personalizes sleep architecture optimization, ensuring deep restorative REM sleep. PSTx stands apart as a promising treatment for chronic insomnia, sleep deprivation, and REM sleep disorders, offering long-term improvement in sleep quality and overall health.
Procedure: Anesthesia-Induced Sleep Therapy — 1. Single-Arm, Non-Randomized Design: All eligible participants receive the same treatment PROSOMNIA Sleep Therapy(PSTx), ensuring consistency and homogeneity.
  2. Targeted Use of Diprivan/Propofol: The PSTx involves the administration of Diprivan/Propofol, an FDA-approved anesthetic, delivered in a controlled environment under the supervision of an Anesthesiologist.
  3. Monitored Anesthesia with Advanced Sleep Assessment: The procedure is monitored according to ASA (American Society of Anesthesiologists) standards, along with real-time EEG to track brain activity during REM sleep.
  4. One (1) Hour PPSTx (60-120 minutes): A PSTx is designed to provide immediate results within a controlled timeframe of 60 to 120 minutes.
  5. Follow-Up Protocol: Post-treatment follow-ups occur at 24 hours, 7 days, and 30 days after the session to measure outcomes and safety parameters.
  6. Focus on Safety and Feasibility: A single-arm approach allows for a concentrated assessment of treatment efficacy.
  Other Names: PROSOMNIA Sleep Therapy; PSTx; PROSOMNIA Sleep
Drug: Diprivan (propofol), Astra-Zeneca — Diprivan/Propofol is a short-acting intravenous anesthetic used in PROSOMNIA Sleep Therapy to induce rapid and controlled REM sleep. Unlike other sleep aids, Propofol works by potentiating GABA_A receptor activity, leading to a deeper and faster transition into sleep. The administration is closely monitored in real-time using EEG to ensure optimal sleep stages are achieved. Propofol is distinct from traditional sedatives due to its precise control, rapid onset, and ability to clear adenosine from the brain, reducing sleep pressure effectively and safely.
  Other Names: Propofol
Device: Continuous EEG Monitoring — Continuous EEG Monitoring is an essential component of PROSOMNIA Sleep Therapy, used to accurately track and optimize sleep architecture in real time. This device provides precise monitoring of brainwave activity, ensuring the patient achieves the necessary stages of REM sleep during therapy. Unlike other monitoring systems, this EEG is used to dynamically adjust the Diprivan/Propofol infusion, allowing for personalized sleep regulation. The continuous data collection helps maintain ideal sleep conditions, distinguishing it from standard sleep therapy interventions that lack real-time neurological insights.
  Other Names: SedLine Brain Function Monitoring; MASIMO SedLine EEG; EEG; SedLine; MASIMO

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of PROSOMNIA Sleep Therapy (PSTx) for individuals suffering from chronic insomnia, sleep deprivation, and REM sleep disorders. Chronic insomnia, characterized by difficulty falling or staying asleep, significantly affects patients and quality of life, mood, and cognitive function. REM sleep disorders, in which the body struggles to enter or maintain restful REM sleep, can worsen these issues. The trial introduces a novel therapy using anesthesia-induced sleep, targeting sleep homeostasis and improving sleep architecture.

Objectives: The primary goals of the trial are to determine:

1. Whether PROSOMNIA Sleep Therapy increases the quality of REM sleep.
2. Whether PSTx increases the duration of REM and/or NREM sleep.
3. Whether PSTx decreases the time it takes participants to fall asleep (sleep onset latency).

Participants will receive ONE (1) PROSOMNIA Sleep Therapy session lasting between 60-120 minutes. Each session uses Diprivan/Propofol to induce sleep, and is monitored via an EEG to ensure proper sleep stages, particularly REM sleep.

Participant Criteria:

Inclusion: Adults aged 18-65 with diagnosed or undiagnosed chronic insomnia or sleep deprivation.

Exclusion: Patients with severe obesity, significant cardiovascular, neurological, or psychiatric conditions, or those with an ASA status above II.

Study Design: This trial is non-randomized, single-arm and open-label, with all participants receiving the PSTx. The trial does not include a comparison group, as the focus is on evaluating the immediate, direct effects of the therapy.

Participants will undergo continuous EEG monitoring during therapy sessions, allowing researchers to track brain activity and sleep stages in real-time. This method ensures that sleep cycles, particularly REM sleep, are optimized for therapeutic benefit.

Therapy Methodology:

PROSOMNIA Sleep Therapy leverages anesthesia to mimic natural sleep patterns and enhance the efficiency of REM sleep. Diprivan/Propofol is used to induce REM sleep, while EEG monitoring tracks and maintains proper sleep architecture throughout the session. The therapy promotes the clearance of adenosine, a compound that builds up during wakefulness and drives the need for sleep. Adenosine is cleared during REM sleep, reducing sleep pressure and improving cognitive function.

Outcome Measures:

Primary Outcomes: Researchers will measure the increase in REM sleep duration, improvement in sleep quality (via self-reported questionnaires), and a reduction in sleep onset latency.

Secondary Outcomes: These include changes in mood, cognitive function, and blood serum uric acid levels. Patient-reported outcomes will also be tracked through tools like the PROSOMNIA Sleep Quiz, which is specifically designed for PSTx.

Significance: Chronic insomnia and REM sleep disorders affect millions globally, leading to cognitive impairment, mood disturbances, and poor overall health. Traditional treatments, including pharmacological approaches and Cognitive Behavioral Therapy for Insomnia (CBT-I), often provide suboptimal results for many individuals. PSTx offers a novel, therapeutic approach to restoring sleep balance and enhancing the overall quality of sleep, particularly for those who have not responded to conventional treatments.

Study Process:

Recruitment and Baseline Assessments: Participants undergo a comprehensive sleep assessment, including sleep questionnaires and polysomnography, to establish a baseline for sleep quality and duration. Blood serum uric acid levels will also be measured to track any biochemical changes due to therapy.

Therapy Sessions: Only one (1) PROSOMNIA Sleep Therapy session will be administered, with the session lasting between 60-120 minutes. Diprivan/Propofol is used to induce sleep, and EEG will monitor brain activity to ensure the proper balance of sleep stages.

Post-Therapy Follow-up: Follow-up assessments will occur at 24 hours, 7 days, and 30 days post-treatment. Researchers will analyze the therapy effects on REM sleep, mood, cognitive function, and other health indicators.

Potential Implications: If successful, this trial could revolutionize how we treat sleep disorders by targeting the underlying mechanisms of sleep pressure and REM sleep disruption. PROSOMNIA Sleep Therapy may offer a safe, effective, and immediate alternative for patients who have exhausted other treatment options.

Key Concepts:

Homeostatic sleep drive, (Process S), caused by adenosine buildup during wakefulness, is disrupted by chronic insomnia. This impacts cognitive function health and recovery. Anesthesia-induced REM sleep via PSTx helps regulate this homeostatic sleep stage, offering deeper and more restorative sleep compared to other sleep therapies. The study uses statistical methods like ANOVA and Chi-square to measure outcomes.

DETAILED DESCRIPTION:
The clinical trial aims to evaluate the safety and efficacy of PROSOMNIA Sleep Therapy (PSTx), an innovative anesthesia-induced treatment, for patients experiencing chronic insomnia, sleep deprivation, and REM sleep disorders. Chronic insomnia, characterized by persistent difficulty falling or staying asleep, often disrupts sleep homeostasis, affecting cognitive function, mood, and overall quality of life. Conventional treatments, such as Cognitive Behavioral Therapy for Insomnia (CBT-I) and pharmacological interventions, frequently yield suboptimal results, making this trial critical for those unresponsive to standard therapies.

Mechanism and Methodology:

PROSOMNIA Sleep Therapy uses a novel approach to target the homeostatic sleep drive by leveraging Diprivan/Propofol, an anesthetic that acts on GABA_A receptors to induce and maintain REM sleep. This process addresses sleep pressure caused by adenosine buildup during wakefulness, promoting its clearance during REM sleep. This controlled anesthesia-induced therapy aims to restore disrupted sleep homeostasis and optimize REM sleep architecture.

During the session, Diprivan/Propofol is administered under Monitored Anesthesia Care (MAC), with continuous EEG monitoring to ensure that sleep stages are appropriately maintained. The single-session therapy, lasting 60-120 minutes, not only aims to enhance REM sleep but also to reduce sleep onset latency (the time required to fall asleep) and improve overall sleep quality.

Study Objectives:

The primary objectives are to determine if PSTx increases REM sleep duration, reduces sleep onset latency, and improves overall sleep quality. Secondary objectives include assessing changes in mood, cognitive function, and biochemical markers (e.g., blood serum uric acid levels).

Broader Implications:

PROSOMNIA Sleep Therapy's innovative method could have broader applications beyond insomnia, including treating mental health disorders (e.g., depression, PTSD), neurodegenerative diseases (e.g., Alzheimer's), and enhancing cardiovascular and metabolic health. Athletes or individuals recovering from injury may also benefit from improved sleep quality and recovery.

Study Design:

This is a non-randomized, single-arm, open-label trial with all participants receiving PSTx to directly observe therapeutic effects without a comparison group. The design allows for focused assessment of therapy outcomes in patients unresponsive to conventional treatments.

Participant Criteria:

Inclusion: Adults aged 18-65 with diagnosed or undiagnosed chronic insomnia or sleep deprivation, with or without prior therapy.

Exclusion: Severe obesity (BMI >35), cardiovascular, neurological, or psychiatric conditions that contraindicate anesthesia, ASA status above II, or diagnosed sleep disorders unrelated to insomnia.

Outcome Measures:

Primary Outcomes: Increased total REM sleep duration (via EEG), improved overall sleep quality (measured by validated questionnaires), and reduced sleep onset latency.

Secondary Outcomes: Changes in cognitive function, mood, and blood serum uric acid levels, tracked through questionnaires and laboratory analyses.

Study Process:

Participants will undergo a comprehensive sleep assessment using polysomnography (PSG) and sleep questionnaires to establish baseline sleep patterns. During the therapy session, Diprivan/Propofol will be administered under anesthesia care, with continuous EEG monitoring to optimize sleep stages. Follow-up assessments at 24 hours, 7 days, and 30 days post-therapy will evaluate changes in REM sleep, mood, cognitive function, and overall health.

Potential Impact:

If successful, this study could position PROSOMNIA Sleep Therapy as a rapid and effective alternative to traditional insomnia treatments, offering hope for individuals unresponsive to current therapies. The study will provide new insights into adenosine clearance, REM sleep regulation, and their roles in cognitive recovery and mood stabilization.

Statistical Analysis:

Primary and Secondary Outcomes: Changes in continuous variables (e.g., REM sleep duration, sleep latency, uric acid levels) will be analyzed using Paired t-tests and ANOVA. Categorical outcomes (e.g., adverse events) will be analyzed using Chi-square tests. Non-normally distributed variables will be evaluated using the Wilcoxon Signed-Rank Test.

Predictive Analysis: Logistic regression will identify baseline variables that predict therapeutic outcomes.

Conclusion:

This trial aims to demonstrate that PROSOMNIA Sleep Therapy can effectively restore sleep homeostasis and improve REM sleep quality, providing a new avenue for treating chronic insomnia and associated conditions. The results could revolutionize the treatment landscape for sleep disorders, particularly in patients who have not found relief with existing options.

The findings will contribute significantly to the field of sleep medicine and open doors for further research in diverse clinical populations, improving sleep health and overall well-being.

ELIGIBILITY:
By adhering to the following criteria, the study aims to select a population that can safely undergo the PROSOMNIA Sleep therapy and for whom the therapy is most likely to be beneficial, ensuring the reliability and validity of the study outcomes.

INCLUSION CRITERIA:

1. Age Range: 18-65 years of age Reason: This age range includes adults who are most likely to benefit from the PROSOMNIA Sleep therapy and who can provide informed consent. It also excludes children and older adults who may have different physiological responses or additional health risks.
2. Diagnosed or Undiagnosed Chronic Insomnia:

   Reason: Included subjects have a consistent pattern of sleep disturbances that PROSOMNIA Sleep Therapy aims to treat.
3. Diagnosed or Undiagnosed Sleep Deprivation:

   Reason: Includes individuals who are not getting enough sleep quantity, which is a key condition that the PROSOMNIA Sleep Therapy aims to address.
4. Diagnosed or Undiagnosed REM Sleep Inconsistencies:

   Reason: Includes individuals who are not getting enough sleep quality and those with specific REM sleep phase issues that the PROSOMNIA Sleep Therapy is designed to improve.
5. Failure to Respond to Conventional Sleep Treatments:

   Reason: Focuses on subjects who have not found relief from existing sleep therapies, ensuring that the study population represents those in need of alternative solutions.
6. Ability to Provide Informed Consent:

Reason: Ensures that participants understand the study and agree to participate voluntarily.

EXCLUSION CRITERIA:

1. Severe Obesity (BMI > 40):

   Reason: Severe obesity can increase the risk of complications with anesthesia and may affect sleep patterns in ways that could confound study results.
2. Cardiovascular Conditions:

   Reason: Patients with significant heart conditions are at higher risk for complications during anesthesia.
3. Neurological Disorders:

   Reason: These diagnosed conditions and medications such as epilepsy could interfere with sleep patterns and responses to sleep therapy.
4. Other Health Conditions Contraindicating Anesthesia:

   Reason: Includes any condition that would make the use of anesthesia unsafe.
5. Greater than ASA II Status:

   Reason: The American Society of Anesthesiologists (ASA) physical status classification system classifies patients based on their pre-anesthesia medical conditions. Excluding those above ASA II ensures that only patients with mild systemic disease are included, to minimize risks.
6. Current Use of Prohibited Medications:

   Reason: Medications that could interfere with the combined use of anesthesia including, but not limited to sedatives and hypnotics; such as benzodiazepines, Z-drugs and barbiturates.
7. Pregnancy or Breastfeeding:

Reason: Ensures the safety of the fetus or infant, as the effects of the PROSOMNIA Sleep therapy on pregnancy or lactation are unknown.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Homeostatic Sleep Pressure | 60-120 minutes
  Evaluate the effectiveness of PROSOMNIA Sleep Therapy in reducing homeostatic sleep pressure, as measured by EEG recordings, blood serum uric acid levels and subjective self-reports.
Change in Sleep Onset Latency | 30 days
  Measure the time it takes for patients to fall asleep (sleep onset latency) following PROSOMNIA Sleep Therapy, using polysomnography (PSG).
Change in REM Sleep Duration | 30 days
  Measure the improvement in the duration of REM sleep using EEG and polysomnography (PSG) before, during and after PROSOMNIA Sleep Therapy.
Change in Overall Sleep Health | 30 days
  The PROSOMNIA Sleep Quiz (PSQ) is a comprehensive tool used to assess sleep health, specifically for identifying chronic insomnia, REM sleep deprivation, or both. The scale measures sleep quality, quantity, and overall health factors contributing to sleep disorders. The PSQ consists of 18 questions, each scoring various sleep and health-related conditions.
  Quiz Scoring System:
  Minimum Score: 0 points Maximum Score: 55 points Higher Scores Indicate: Poorer sleep health and worse outcomes.

SECONDARY OUTCOMES:
Changes in Blood Serum Uric Acid Levels | 60-120 minutes
  Measure changes in blood serum uric acid levels, reflecting adenosine release into the bloodstream, after PROSOMNIA Sleep Therapy sessions.
Improvement in Patient-Reported Mood | 30 days
  The Mood Quality Assessment is used to evaluate the impact of PROSOMNIA Sleep Therapy on patient-reported mood following treatment. This assessment utilizes a 5-point scale:
  Minimum Value: 1 (Happy) Maximum Value: 5 (Bad) Higher scores indicate worse mood outcomes, reflecting increased mood disturbances or negative emotional states. The assessment is conducted at baseline and post-treatment to gauge changes in mood and emotional well-being, providing insights into the therapy's effect on overall mood regulation and mental health.

OTHER OUTCOMES:
Adverse Event Reporting | 6 months
  Record any adverse events associated with PROSOMNIA Sleep Therapy, categorized by severity and likelihood of relation to the intervention.
PROSOMNIA Sleep Virtual Consultation Note | 30 days
  The data collected during the PROSOMNIA Sleep Virtual Consultation Note will establish baseline characteristics, identify risks and create a Personalized PROSOMNIA Sleep Therapy Plan. This plan will integrate specific interventions to address risk factors and enhance treatment effectiveness. Continuous monitoring and periodic reassessment will be conducted to identify any emerging patterns, modify interventions as needed, and ensure long-term improvements in sleep health and overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Nyree Penn, MHSc., CAA, Master of Health Science, Principal Investigator — Memorial Healthcare System
Locations (1):
- PROSOMNIA Sleep Health and Wellness, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share individual participant data (IPD) that underlie the results presented in any forthcoming publications resulting from this trial. This includes all IPD collected and used for analysis and publication, such as de-identified data sets related to primary and secondary outcome measures, baseline characteristics, and adverse event reports. The data will be made available to researchers upon request to promote transparency, reproducibility, and further exploration of the study's findings. Access will be granted in accordance with ethical guidelines and data-sharing policies to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The individual participant data (IPD) and supporting information will be available starting 6 months after the publication of the primary study results. The data will remain accessible for 5 years following the initial release. After this period, access may be reviewed and extended upon request.
Access Criteria: The individual participant data (IPD) and supporting information will be accessible to qualified researchers affiliated with academic institutions, healthcare organizations, or industry partners involved in sleep medicine research. Researchers must submit a detailed research proposal outlining the purpose and objectives of their study.
  Access will be granted following approval by an independent review board to ensure the scientific merit and ethical use of the data. Researchers will be required to sign a data use agreement (DUA) to maintain confidentiality and adhere to ethical guidelines. Data will be shared through a secure online platform.
URL: https://drive.google.com/file/d/1ChQlpKLVuhUMWeQNxl-IAfwJ1jHEg8b2/view

REFERENCES:
- [Background] Saito H, Nishimura M, Shibuya E, Makita H, Tsujino I, Miyamoto K, Kawakami Y. Tissue hypoxia in sleep apnea syndrome assessed by uric acid and adenosine. Chest. 2002 Nov;122(5):1686-94. doi: 10.1378/chest.122.5.1686. PMID 12426272
- [Background] Hirotsu C, Tufik S, Guindalini C, Mazzotti DR, Bittencourt LR, Andersen ML. Association between uric acid levels and obstructive sleep apnea syndrome in a large epidemiological sample. PLoS One. 2013 Jun 24;8(6):e66891. doi: 10.1371/journal.pone.0066891. Print 2013. PMID 23826169
- [Background] Korkutata M, Lazarus M. Adenosine A2A receptors and sleep. Int Rev Neurobiol. 2023;170:155-178. doi: 10.1016/bs.irn.2023.04.007. Epub 2023 Apr 29. PMID 37741690
- [Background] Lazarus M, Chen JF, Huang ZL, Urade Y, Fredholm BB. Adenosine and Sleep. Handb Exp Pharmacol. 2019;253:359-381. doi: 10.1007/164_2017_36. PMID 28646346
- [Background] Murdock MH, Yang CY, Sun N, Pao PC, Blanco-Duque C, Kahn MC, Kim T, Lavoie NS, Victor MB, Islam MR, Galiana F, Leary N, Wang S, Bubnys A, Ma E, Akay LA, Sneve M, Qian Y, Lai C, McCarthy MM, Kopell N, Kellis M, Piatkevich KD, Boyden ES, Tsai LH. Multisensory gamma stimulation promotes glymphatic clearance of amyloid. Nature. 2024 Mar;627(8002):149-156. doi: 10.1038/s41586-024-07132-6. Epub 2024 Feb 28. PMID 38418876
- [Background] Nelson LE, Franks NP, Maze M. Rested and refreshed after anesthesia? Overlapping neurobiologic mechanisms of sleep and anesthesia. Anesthesiology. 2004 Jun;100(6):1341-2. doi: 10.1097/00000542-200406000-00003. No abstract available. PMID 15166550
- [Background] Tung A, Bergmann BM, Herrera S, Cao D, Mendelson WB. Recovery from sleep deprivation occurs during propofol anesthesia. Anesthesiology. 2004 Jun;100(6):1419-26. doi: 10.1097/00000542-200406000-00014. PMID 15166561
- [Background] Vacas S, Kurien P, Maze M. Sleep and Anesthesia - Common mechanisms of action. Sleep Med Clin. 2013 Mar;8(1):1-9. doi: 10.1016/j.jsmc.2012.11.009. No abstract available. PMID 28747855
- [Background] Eleveld DJ, Colin P, Absalom AR, Struys MMRF. Pharmacokinetic-pharmacodynamic model for propofol for broad application in anaesthesia and sedation. Br J Anaesth. 2018 May;120(5):942-959. doi: 10.1016/j.bja.2018.01.018. Epub 2018 Mar 12. PMID 29661412
- [Background] Murphy M, Bruno MA, Riedner BA, Boveroux P, Noirhomme Q, Landsness EC, Brichant JF, Phillips C, Massimini M, Laureys S, Tononi G, Boly M. Propofol anesthesia and sleep: a high-density EEG study. Sleep. 2011 Mar 1;34(3):283-91A. doi: 10.1093/sleep/34.3.283. PMID 21358845
- [Background] Yang CM, Lin SC, Cheng CP. Transient insomnia versus chronic insomnia: a comparison study of sleep-related psychological/behavioral characteristics. J Clin Psychol. 2013 Oct;69(10):1094-107. doi: 10.1002/jclp.22000. Epub 2013 Jun 24. PMID 23797824
- [Background] Siegel JM. The neurotransmitters of sleep. J Clin Psychiatry. 2004;65 Suppl 16(Suppl 16):4-7. PMID 15575797
- [Background] Vyazovskiy VV. Sleep, recovery, and metaregulation: explaining the benefits of sleep. Nat Sci Sleep. 2015 Dec 17;7:171-84. doi: 10.2147/NSS.S54036. eCollection 2015. PMID 26719733
- [Background] Roth T, Roehrs T, Pies R. Insomnia: pathophysiology and implications for treatment. Sleep Med Rev. 2007 Feb;11(1):71-9. doi: 10.1016/j.smrv.2006.06.002. Epub 2006 Dec 18. PMID 17175184
- [Background] Xu Z, Jiang X, Li W, Gao D, Li X, Liu J. Propofol-induced sleep: efficacy and safety in patients with refractory chronic primary insomnia. Cell Biochem Biophys. 2011 Jul;60(3):161-6. doi: 10.1007/s12013-010-9135-7. PMID 21107748
- See also: Welcome to the PROSOMNIA Sleep Clinical Trials information page! Here, potential participants can learn more about our innovative clinical research dedicated to advancing sleep health and wellness — https://prosomniasleep.com/m/login?r=%2Fclinical-trials
- See also: PROSOMNIA Sleep Health &amp;amp; Wellness is dedicated to revolutionizing sleep health through innovative therapies and solutions. The website provides information on cutting-edge sleep therapies, including anesthesia-induced treatments. — https://prosomniasleep.com/
- Available data/document: Statistical Analysis Plan: PSHW Statistical Analysis Plan — https://drive.google.com/file/d/1iSQ5KoBNJtChtg1vSJDVFlar7D8ntaxI/view?usp=sharing — Study Protocol and Statistical Analysis Plan (SAP)
- Available data/document: Individual Participant Data Set: Virtual Consultation SOAP Note — https://drive.google.com/file/d/1uAAbC0gRFOthwnUiWz3O2sDyLgkGkiKf/view?usp=sharing — Virtual Consultation SOAP Note
- Available data/document: Informed Consent Form: PSHW Informed Consent — https://docs.google.com/document/d/1Otiwf8P6Rozk_MyA5qDgCnx-J7lXfJsfm0He5j5U9_I/edit?usp=sharing — PSHW Informed Consent For Research
- Available data/document: Individual Participant Data Set: PROSOMNIA Sleep Quiz — https://drive.google.com/file/d/1XWzVYL0L2OR8FzFUGtd0vggjwBflBAFa/view?usp=sharing — PROSOMNIA Sleep Quiz
- Available data/document: Clinical Study Report: Sleep Quiz Evaluation — https://drive.google.com/file/d/1Hzw1OvpbAn44nCbvqbtPwC25clwCbclW/view?usp=sharing — PSHES Sleep Quiz Scoring System
- Available data/document: Individual Participant Data Set: Mood/Emotion Quality Scale — https://drive.google.com/file/d/1-UzkVbn7UG57aZMg9d1LRB9yoLkjUlWS/view?usp=sharing — Mood/Emotion Quality Scale